CLINICAL TRIAL: NCT04528810
Title: A Prospective Observational Study of Child Injury Based on Data Mining
Brief Title: A Study of Child Injury Based on Data Mining
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFU20200816
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Injuries; Child
Keywords: Injuries; Child; Epidemiology
MeSH Terms: conditions — Wounds and Injuries | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Child injuries: pediatric patients under the age of 18 years newly diagnosed with injuries in the emergency department
  Interventions: Other: not applicable (Observational Study)

INTERVENTIONS:
Other: not applicable (Observational Study) — This is an observational study and does not include interventions.

SUMMARY:
A comprehensive pediatric injury burden assessment is an essential foundation for formulating injury prevention strategies and improving emergency care for injured children. Although the hospital-based passive surveillance of national injury surveillance system of medical and health institutions has been well-established in China, the monitoring points of hospitals were not stratified according to children's hospital. Aim of the project is to collect epidemiological and clinical data to describe causes, clinical features and outcomes of pediatric injuries at a Children's Hospital in Shanghai, China. The project intends to establish a method for collecting and analyzing high quality data of child injury using data mining based on the hospital information system.

DETAILED DESCRIPTION:
Injuries are a leading cause of death for infants and children around the world. According to the Haddon Injury Control Model, 90 percent of injuries are both predictable and preventable. Injuries are preventable, not "accidents". All unintentionally and intentionally injured children first visit to the emergency department are recruited in the study. Children's Hospital of Fudan University with a Regional Pediatric Trauma Centre is also the first Pediatric Injury Prevention Center established in China. We conduct a prospective cohort study to investigate the epidemiology, clinical course, and outcomes of the injured child first visit to the emergency department, which expected to serve as evidence of injury prevention and promising practices. In the study, we collect and analyze high quality data of child injury based on data mining.

ELIGIBILITY:
Inclusion Criteria:

All pediatric patients between the ages of 0-18 years newly diagnosed with injuries in the emergency department，and recorded ICD-10 diagnosis codes from V01 to X39

Exclusion Criteria:

Patients who were dead on arrival to the emergency department are not included.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients between the ages of 0-18 years newly diagnosed with injuries
Sampling Method: Probability Sample
Enrollment: 10762 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of injury categories | At baseline
  According to the electronic medical record system, the distribution of injury categories is defined as the proportion of various injury causes (fall，motor vehicle crash，sports, struck, foreign body) in the cohort subjects.

SECONDARY OUTCOMES:
28 days mortality | Within 28 days from ED admission
  Mortality within 28 days from Emergency Department（ED）admission based on electronic medical records system
180 days mortality | Within 180 days from ED admission
  Mortality based on electronic medical records system
Short-term disability | At 180 days from ED admission
  Disability accessed by the Glasgow Outcome Scale (GOS) at 180 days from ED admission. The Glasgow Outcome Scale was dichotomized into favorable outcome (moderate disability or good recovery ; GOS score of 4 or 5) and unfavorable outcome (death, vegetative state or severe disability; GOS score 1-3).
Percentage of ICU admission | From ED admission to 72 hours
  Percentage of ICU admission from ED admission to 72 hours based on electronic medical records system

IPD SHARING:
Plan to Share IPD: Undecided